CLINICAL TRIAL: NCT06079060
Title: A Functional Performance and Acceptability Evaluation of Synthetic Nitrile Male Condom Compared to a Standard Latex Male Condom
Brief Title: Evaluation of Synthetic Nitrile Male Condom Compared to Standard Latex Male Condom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karex Industries Sdn. Bhd. (Industry)
Collaborators: Match Research (Other); Essential Access Health (Other); Sigma3 Services SARL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Karex03
Record Dates: First submitted 2023-09-20; First posted 2023-10-12 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Sexually Transmitted Diseases
Keywords: Synthetic Male Condom; Slippage-Breakage Study
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: A sequential randomised 2-period cross-over trial comparing five uses of a 61 mm width synthetic nitrile male condom with five uses of a 61 mm width standard latex male condom.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each product will be labeled with a randomly generated code.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Synthetic Nitrile Condom (61mm) (Experimental): 61mm width synthetic Nitrile condoms
  Interventions: Device: Synthetic Nitrile Condom (61mm)
- Control Latex Condom (Active Comparator): 61mm width Natural Rubber Latex condoms
  Interventions: Device: Control Latex Condom

INTERVENTIONS:
Device: Synthetic Nitrile Condom (61mm) — 61mm width Synthetic Nitrile Condoms
  Arms: Synthetic Nitrile Condom (61mm)
Device: Control Latex Condom — 61mm width Natural Rubber Latex Condom
  Arms: Control Latex Condom

SUMMARY:
Thia is a multi-site, randomised 2-period cross-over trial comparing five uses of a 61 mm width synthetic nitrile male condom with five uses of a 61 mm width standard latex male condom.

DETAILED DESCRIPTION:
A sequential randomised 2-period cross-over trial comparing five uses of a 61 mm width synthetic nitrile male condom with five uses of a 61 mm width standard latex male condom. Each couple will be asked to use five synthetic nitrile condoms, and five latex control male condoms in a randomised order. Couples will complete a Condom Use Report after each condom use. Function, safety, and acceptability will be assessed at each of two follow-up visits conducted after using each set of five condoms. The trial will enrol up to 300 couples, anticipating that at least 255 couples will complete the study. Half of the couples (150) will be enrolled in Durban, South Africa and half (150) enrolled in California USA.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 45 years (inclusive);
2. Be literate (able to read a newspaper or letter easily);
3. Have been in an exclusive (monogamous) sexual relationship with partner for at least 3 months; and intend to continue to be an exclusive (monogamous) sexual relationship with their spouse or partner while participating in this research study;
4. Be sexually active (defined as having at least one vaginal coital act per week);
5. Willing to give informed consent;
6. Willing to complete the male condom coital use reports;
7. Willing to use the study condoms as directed;
8. Agree to use only the study lubricant provided;
9. Agree to only use the study condoms sequentially during time of participation
10. Willing to adhere to the follow-up schedule and all study procedures;
11. Willing to provide research study staff with an address, phone number or other locator information while participating in the study;
12. Willing to participate in the study for the duration of 10 condom uses (approximately 2-3 months);
13. Willing to provide photo identification and/or have fingerprint scan to exclude co-enrolment in other research projects;
14. Female partner using hormonal or other non-barrier contraception (e.g. OCs, injectable, implant, Intrauterine device (IUD), or have had a tubal sterilization) or male partner vasectomised;
15. Agree to return any unopened condoms;
16. Male partner willing to ejaculate during vaginal intercourse;
17. Male partner willing to hold on to the condom ring when withdrawing the erect penis after sexual intercourse;
18. Agree to not bring study condoms in contact with genital or oral piercing jewelry
19. EAH: Both partners have valid personal email and operable mobile phones;
20. Former participant in Karex02 Study: male partner measures at least 118 mm in girth of erect penis.
21. Agree that information provided in Karex02 study may be used and combined with the information in this study

Exclusion Criteria:

1. Female partner is pregnant or desires to become pregnant during the time of the research study;
2. Either partner is known to be HIV positive (based on self report [EAH] or documented HIV-negative test result within past two months;
3. Self-reported history of recurrent sexually transmitted infection (e.g. gonorrhea, syphilis, Chlamydia);
4. Male partner has known erectile or ejaculatory dysfunction;
5. Either partner has genital piercing jewelry, uses genital beading or uses sex toys, drugs, medications or non-study devices that can affect sexual performance;
6. Either partner has known sensitivities or allergies to latex, synthetic nitrile, vaginal/sexual lubricants or lubricants used on condoms;
7. Either partner reports symptoms of STI (EAH) or has observable evidence of STI as determined through syndromic diagnosis and vaginal/penile examination (MRU);
8. Either partner is currently participating in another condom study;
9. Either partner is a past or current employee of Essential Access Health, University of the Witwatersrand, or Karex;
10. Either partner is a sex worker.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 305 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Clinical breakage | 3 - 5 months
  Clinical breakage is defined as breakage or tearing during sexual intercourse or during withdrawal of the male condom from the vagina. Clinical breakage is breakage with potential adverse clinical consequences. The clinical breakage rate is calculated by dividing the number of male condoms reported to have broken or torn during sexual intercourse or during withdrawal by the number of male condoms used during vaginal intercourse.
Clinical slippage | 3 - 5 months
  Clinical slippage is defined as a condom slipping completely off the penis during sexual intercourse or during withdrawal from the vagina. The clinical slippage rate is calculated by dividing the number of male condoms that slipped by the number of male condoms used during vaginal intercourse.
Clinical failure | 3 - 5 months
  Clinical failure is defined as a clinical breakage or a clinical slippage. The clinical failure rate is calculated by dividing the number of male condoms with a clinical failure by the number of male condoms used during vaginal intercourse.

SECONDARY OUTCOMES:
Genital discomfort | 3 - 5 months
  Rates of genital discomfort reported to have occurred during or immediately after condom use. Genital adverse events will be classified by relatedness, expectedness and severity.
Acceptability i.e Comfort in use, ease of fitting and removal, like or dislike of product attributes, adequacy and feel of lubrication. | 3 - 5 months
  Questionnaires obtained after participants complete 5 condom uses of each condom type cover multiple acceptability factors. For these acceptability measures, Likert scores ranging from 1 (lowest) to 5 (highest) will be compared across condom types.
Non-Clinical breakage | 3 - 5 months
  Defined as breakage noticed before sexual intercourse or occurring after withdrawal of the male condom from the vagina. Non-clinical breakage is breakage with no potential adverse clinical consequences. The non-clinical breakage rate is calculated by dividing the number of male condoms reported to have broken before sexual intercourse or after withdrawal by the number of male condom packages opened.
Non-Clinical slippage | 3 - 5 months
  Defined as slippage along the shaft of the penis during sexual intercourse (but not completely off the penis). Non-clinical slippage is slippage with no potential adverse clinical consequences. The non-clinical slippage rate is calculated by dividing the number of male condoms reported to have partially slipped during sexual intercourse by the number of male condoms used during vaginal intercourse.

CONTACTS AND LOCATIONS:
Overall Officials: Mags Beksinska, PhD, Principal Investigator — MRU (MatCH Research Unit)
Locations (3):
- United States (2):
  - Essential Access Health, Berkeley, California
  - Essential Access Health, Los Angeles, California
- MRU (MatCH Research Unit), Durban, South Africa

IPD SHARING:
Plan to Share IPD: No